CLINICAL TRIAL: NCT03087591
Title: Safety and Immunologic Activity of Multiple Infusions of APN401
Brief Title: APN401 in Treating Patients With Recurrent or Metastatic Pancreatic Cancer, Colorectal Cancer, or Other Solid Tumors That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00041173; NCI-2017-00050 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 03716 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2017-01-13; First posted 2017-03-22 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: Metastatic Malignant Neoplasm in the Brain; Metastatic Solid Neoplasm; Recurrent Colorectal Carcinoma; Recurrent Pancreatic Carcinoma; Recurrent Solid Neoplasm; Stage IV Colorectal Cancer; Stage IV Pancreatic Cancer; Stage IVA Colorectal Cancer; Stage IVA Pancreatic Cancer; Stage IVB Colorectal Cancer; Stage IVB Pancreatic Cancer; Unresectable Solid Neoplasm
MeSH Terms: conditions — Brain Neoplasms; Neoplasm Metastasis; Colorectal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (APN401) (Experimental): Patients receive siRNA-transfected peripheral blood mononuclear cells APN401 IV over 30 minutes on days 1, 29, and 57 in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: siRNA-transfected Peripheral Blood Mononuclear Cells (PBMC) APN401

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: siRNA-transfected Peripheral Blood Mononuclear Cells (PBMC) APN401 — Given IV
  Other Names: APN401; siRNA-transfected PBMC APN401

SUMMARY:
This phase I trial studies the side effects and best dose of APN401 in treating patients with pancreatic cancer, colorectal cancer, or other solid tumors that have spread to other places in the body or have come back. APN401 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities and establish the safety of multiple infusions of small interfering ribonucleic acid (siRNA)-transfected peripheral blood mononuclear cells APN401 (APN401).

SECONDARY OBJECTIVES:

I. To determine the immunologic effects of multiple infusions of APN401. II. To document clinical response and survival.

OUTLINE:

Patients receive siRNA-transfected peripheral blood mononuclear cells APN401 intravenously (IV) over 30 minutes on days 1, 29, and 57 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed inoperable, recurrent or metastatic malignant solid tumors, deemed incurable, and who have either:

  * Failed to respond to standard therapy or
  * For whom no standard therapy is available or
  * Refuse to receive standard therapies
* The study is intended to enroll patients with pancreatic and colorectal cancer; patients with other types of solid tumors will require approval by the principal investigator
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
* Patients with treated, stable, and asymptomatic brain metastases are eligible
* Patients on every 3 or every 4 week systemic therapy programs must be at least 4 weeks since treatment and recovered from any clinically significant toxicity experienced; patients on weekly or daily systemic therapy programs and patients receiving radiation must be at least 1 week since treatment and recovered from any clinically significant toxicity experienced; must be at least 4 weeks and have recovered from major surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* White blood cells >= 3000/uL
* Platelets >= 100,000/uL
* Hematocrit >= 28%
* Creatinine =< 1.6 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal
* Bilirubin =< 1.6 mg/dL (except patients with Gilbert's syndrome, who must have a total bilirubin less than 3.0 mg/dL)
* Albumin >= 3.0 g/dL
* International normalized ratio (INR) =< 1.5

Exclusion Criteria:

* Women must not be pregnant or breastfeeding; all women of childbearing potential must have a blood test within 72 hours to rule out pregnancy; women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception; women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for 26 weeks after the last dose of investigational product, in such a manner that the risk of pregnancy is minimized; sexually mature females who have not undergone a hysterectomy or who have not been postmenopausal naturally for at least 24 consecutive months (i.e., who have had menses at some time in the preceding 24 consecutive months) are considered to be of childbearing potential; women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential
* Untreated, progressing, or symptomatic brain metastases
* Autoimmune disease, as follows: patients with a history of inflammatory bowel disease are excluded as are patients with a history of symptomatic disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]); patients with motor neuropathy considered of autoimmune origin (e.g., Guillain-Barre syndrome and myasthenia gravis) are excluded; patients with a history of autoimmune thyroiditis are eligible if their current thyroid disorder is treated and stable with replacement or other medical therapy
* Any other malignancy from which the patient has been disease-free for less than 2 years, with the exception of adequately treated and cured basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Other ongoing systemic therapy for cancer, including any other experimental treatment; these include concomitant therapy with any of the following: IL-2, interferon, ipilimumab, pembrolizumab, nivolumab, or other immunotherapy; cytotoxic chemotherapy; and targeted therapies
* Ongoing requirement for an immunosuppressive treatment, including the use of glucocorticoids or cyclosporine, or with a history of chronic use of any such medication within the last 4 weeks before enrollment; patients are excluded if they have any concurrent medical condition that requires the use of systemic steroids (the use of inhaled or topical steroids is permitted)
* Infection with human immunodeficiency virus (HIV)
* Active infection with hepatitis B; active or chronic infection with hepatitis C
* Clinically significant pulmonary dysfunction, as determined by medical history and physical examination; patients with a history of pulmonary dysfunction must have pulmonary function tests with a forced expiratory volume in 1 second (FEV1) >= 60% of predicted and a diffusing capacity of the lung for carbon monoxide (DLCO) >= 55% (corrected for hemoglobin)
* Clinically significant cardiovascular abnormalities (e.g., congestive heart failure or symptoms of coronary artery disease), as determined by medical history and physical examination; patients with a history of cardiac disease must have a normal cardiac stress test (treadmill, echocardiogram, or myocardial perfusion scan) within the past 6 months of study entry
* Active infections or oral temperature > 38.2 degrees Celsius (C) within 48 hours of study entry
* Systemic infection requiring chronic maintenance or suppressive therapy
* Patients are excluded for any underlying medical or psychiatric condition, which in the opinion of the investigator, will make treatment hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent rashes or diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Triozzi, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Wolf D, Baier G. IFNgamma Helps CBLB-Deficient CD8+ T Cells to Put Up Resistance to Tregs. Cancer Immunol Res. 2022 Apr 1;10(4):370. doi: 10.1158/2326-6066.CIR-22-0080. PMID 35362047

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (APN401): Patients receive siRNA-transfected peripheral blood mononuclear cells APN401 IV over 30 minutes on days 1, 29, and 57 in the absence of disease progression or unacceptable toxicity.
  Laboratory Biomarker Analysis: Correlative studies
  siRNA-transfected Peripheral Blood Mononuclear Cells APN401: Given IV
Period: Overall Study
Arm/Group | Treatment (APN401)
Started | 11
Completed | 9
Not Completed | 2
Not completed — Disease progression before starting treatment, removed from study | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Out of the 11 participants, only 9 actually received treatment have data collected.
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 56 [36 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
CD3+ [Mean (Standard Deviation); unit: percentage of cells] | 27.4 (16.4)
CD4+ [Mean (Standard Deviation); unit: percentage of cells] | 24.2 (26.8)
CD8+ [Mean (Standard Deviation); unit: percentage of cells] | 19.3 (23.7)
CD4+ICOS+ [Mean (Standard Deviation); unit: percentage of cells] | 13.2 (20.0)
CD8+ICOS+ [Mean (Standard Deviation); unit: percentage of cells] | 11.3 (14.2)
CD4+FOXP3+ [Mean (Standard Deviation); unit: percentage of cells] | 12.0 (14.7)
CD4+CD45RO+ [Mean (Standard Deviation); unit: percentage of cells] | 26.2 (19.2)
CD3-CD56+ [Mean (Standard Deviation); unit: percentage of cells] | 4.2 (2.8)
CD14+ [Mean (Standard Deviation); unit: percentage of cells] | 6.0 (6.6)
CD19+ [Mean (Standard Deviation); unit: percentage of cells] | 2.6 (4.9)
CD56+ [Mean (Standard Deviation); unit: percentage of cells] | 4.9 (4.2)
Neutrophil to Lymphocyte Ratio [Mean (Standard Deviation); unit: ratio] | 3.32 (1.20)
IFN [Mean (Standard Deviation); unit: pg/ml] | 65.1 (17.7)
IL-2 [Mean (Standard Deviation); unit: pg/ml] | 195.1 (231.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events Common Terminology Criteria for Adverse Events Version 4.0
Description: Will be categorized by organ system and severity, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events. Related treatment emergent adverse events by maximum severity. Unexpected grade 4 and all grade 5 events are considered severe adverse events.
  CTCAE grades 3-5 allergic reactions related to study cell infusion CTCAE grades 3 and greater autoimmune reactions other than that vitiligo CTCAE grades 3 and greater organ toxicity (cardiac, dermatologic, gastrointestinal, hepatic, pulmonary, renal/genitourinary or neurologic) not pre-existing or due to the underlying malignancy and occurring within 30 days of study product infusion
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
Participants
  General disorders and administration site conditions: Unobserved | 0
  General disorders and administration site conditions: Grade 1 | 1
  General disorders and administration site conditions: Grade 2 | 8
  General disorders and administration site conditions: Grade 3 | 0
  Nervous System Disorders: Unobserved | 5
  Nervous System Disorders: Grade 1 | 4
  Nervous System Disorders: Grade 2 | 0
  Nervous System Disorders: Grade 3 | 0
  Gastrointestinal Disorders: Unobserved | 6
  Gastrointestinal Disorders: Grade 1 | 2
  Gastrointestinal Disorders: Grade 2 | 0
  Gastrointestinal Disorders: Grade 3 | 1
  Musculoskeletal and connective tissue disorders: Unobserved | 7
  Musculoskeletal and connective tissue disorders: Grade 1 | 0
  Musculoskeletal and connective tissue disorders: Grade 2 | 2
  Musculoskeletal and connective tissue disorders: Grade 3 | 0

2. Secondary Outcome: Clinical Response as Assessed by RECIST
Description: Will be summarized as frequency counts and percentages. RECIST criteria: Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD; Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Up to approximately 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 3
  Progressive Disease | 6

3. Secondary Outcome: Frequency of Immune Cells
Description: Immune response as measured by frequency of immune cells
Time Frame: Days 15 and 28
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
percentage of cells
  CD3+ (day 15) | 37.1 (17.3)
  CD3+ (day 28) | 40.3 (15.1)
  CD4+ (day 15) | 19.0 (20.0)
  CD4+ (day 28) | 26.4 (4.0)
  CD8+ (day 15) | 15.5 (16.1)
  CD8+ (day 28) | 22.7 (14.1)
  CD14+ (day 15) | 5.1 (2.8)
  CD14+ (day 28) | 7.3 (7.3)
  CD19+ (day 15) | 1.2 (1.6)
  CD19+ (day 28) | 2.6 (3.2)
  CD45RO+ (day 15) | 14.8 (8.2)
  CD45RO+ (day 28) | 37.3 (2.0)
  CD56+ (day 15) | 4.8 (3.4)
  CD56+ (day 28) | 8.3 (8.5)
  CD4+ICOS+ (day 15) | 12.8 (19.7)
  CD4+ICOS+ (day 28) | 16.8 (15.7)
  CD4+CD45RO+ (day 15) | 14.8 (8.2)
  CD4+CD45RO+ (day 28) | 37.3 (2.0)
  CD4+FOXP3+ (day 15) | 13.9 (16.4)
  CD4+FOXP3+ (day 28) | 29.5 (18.3)
  CD8+ICOS+ (day 15) | 12.3 (14.5)
  CD8+ICOS+ (day 28) | 25.2 (7.8)
  CD3-CD56+ (day 15) | 4.2 (1.7)
  CD3-CD56+ (day 28) | 5.4 (1.1)

4. Secondary Outcome: Immune Response as Measured by Interferon Production
Description: Immune response as measured by interferon production
Time Frame: Days 15 and 28
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
pg/ml
  IFN (day 15) | 75.1 (17.6)
  IFN (day 28) | 90.7 (37.8)
  IL-2 (day 15) | 226 (51.1)
  IL-2 (day 28) | 674.4 (978.6)

5. Secondary Outcome: Neutrophil to Lymphocyte Ratio
Description: Immune response as measured by neutrophil to lymphocyte ratio
Time Frame: Days 15 and 28
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
ratio
  Day 15 | 2.72 (1.21)
  Day 28 | 4.98 (5.81)

6. Secondary Outcome: Overall Survival (OS)
Description: Exploratory survival plots will be estimated using the Kaplan Meier approach and median overall survival will be estimated if enough events occur.
Time Frame: From the initial infusion to confirmation of death, assessed up to approximately 4 years
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
days | 181 [47 to 707]

7. Secondary Outcome: Progression-free Survival (PFS)
Description: Exploratory survival plots will be estimated using the Kaplan Meier approach and median PFS will be estimated if enough events occur.
Time Frame: From the initial infusion to confirmation of progression or death, assessed up to approximately 4 years
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (APN401)
Number analyzed (Participants) | 9
days | 70 [47 to 237]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during treatment and follow up 30 days past treatment and up to approximately 4 years for survival.
Arm/Group | Treatment (APN401)
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (APN401) (N=9)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ASCITES (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
FATIGUE (General disorders) | 1 (1)
HEPATIC HEMORRHAGE (Hepatobiliary disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (APN401) (N=9)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (4)
ASCITES (Gastrointestinal disorders) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (7)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (2)
CHILLS (General disorders) | 8 (21)
EDEMA LIMBS (General disorders) | 1 (1)
FATIGUE (General disorders) | 4 (4)
FEVER (General disorders) | 3 (5)
FLU LIKE SYMPTOMS (General disorders) | 1 (1)
RIGORS (General disorders) | 1 (2)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
ALKALINE PHOSPHATASE INCREASE (Investigations) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BLOOD BILIRUBIN INCREASE (Investigations) | 2 (2)
CREATININE INCREASE (Investigations) | 1 (2)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (3)
HYPERURICEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 2 (4)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (2)
HYPONATREMIA (Metabolism and nutrition disorders) | 2 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
BACK SPASM (Musculoskeletal and connective tissue disorders) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (2)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (3)
HEADACHE (Nervous system disorders) | 5 (14)
PARESTHESIA (Nervous system disorders) | 2 (2)
CYSTITIS NONINFECTIVE (Renal and urinary disorders) | 1 (1)
DYSURIA (Renal and urinary disorders) | 1 (1)
HEMATOMA (Vascular disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT03087591/Prot_SAP_001.pdf
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03087591/ICF_000.pdf